CLINICAL TRIAL: NCT02744014
Title: Evidence-Based Mindset & Physical Therapy for Add-on Treatment of Active Axial Spondyloarthritis: Safety and Efficacy
Brief Title: Add-on Therapy for Axial Spondyloarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Bernhoven Hospital (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, D.L.P. Baeten, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Academic_Medical_Center
Record Dates: First submitted 2016-03-02; First posted 2016-04-19 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early intervention group (Experimental): The program starts with a 30-days training course led by course instructor Wim Hof and supervised by the research team. The mindset & physical therapy based on the Wim Hof Method includes breathing techniques, training of mindset and concentration, and gradual cold exposure.
  Interventions: Behavioral: Add-on Therapy for Axial Spondyloarthritis
- Late intervention group (Other): This group will receive the same training with a delay of 60-90 days, serving initially as control.
  Interventions: Behavioral: Add-on Therapy for Axial Spondyloarthritis

INTERVENTIONS:
Behavioral: Add-on Therapy for Axial Spondyloarthritis
  Other Names: Wim Hof Method

SUMMARY:
Rationale: Recent investigations suggest that, through certain concentration/meditation techniques, it is possible to modulate autonomic activity. The results of a recent randomized controlled trial investigating the "Wim Hof Method" have shown a direct biological effect on in-vivo cytokine production and are strongly encouraging the clinical evaluation of the technique's efficacy in immune-mediated inflammatory diseases.

Objective: To investigate whether an add-on mindset & physical therapy program based on the "Wim Hof Method" can safely and efficaciously be applied in patients with active axial spondyloarthritis.

Study design: Prospective open-label randomized controlled trial, safety and efficacy.

Study population: Twenty-four patients with active axial spondyloarthritis between 18 and 45 years of age.

Intervention: A 30-day training program of add-on mindset and physical therapy for axial spondyloarthritis, using the methodology as designed and instructed by Wim Hof. It involves breathing techniques, training of mindset and concentration, and gradual cold exposure.

Main study parameters/endpoints: Safety evaluation of the program is the primary aim of the study. Secondary endpoint is the modulation of serum CRP levels. Exploratory objectives include modulation of clinical disease activity (ASDAS), quality of life (SF-36, EQ-5D), depressive symptoms (HADS), and predictive role of generalized and specific outcome expectancies (EPQ-N, LOT-R, VAS scales).

DETAILED DESCRIPTION:
Axial spondyloarthritis (axSpA) is a common systemic autoinflammatory disease affecting approximately 7 in 1.000 individuals. Recent investigations suggest that, through certain concentration/meditation techniques, it is possible to modulate autonomic activity. The endotoxemia experiment in an individual (named Wim Hof) who used a self-created concentration/meditation technique is strongly supportive of these findings. The use of his technique - including breathing techniques, training of mindset and concentration, and gradual cold exposure - seemed to evoke a controlled stress response. This response was characterized by sympathetic nervous system activation and subsequent catecholamine/cortisol release, which seemed to attenuate the innate immune response. The remarkable results in the studied individual led to a randomised controlled trial of this technique at the Radboud UMC. Twenty-four healthy individuals were randomised to receive an instruction course of the technique or no instructions at all and subsequently underwent an endotoxemia experiment. The experiment involved the intravenous administration of very low doses of lipopolysaccharide and measuring the in-vivo cytokine response and clinical symptoms. The results of this study have shown a direct biological effect on in-vivo cytokine production and are strongly encouraging the evaluation of the technique's efficacy in clinical practice.

The techniques of the Wim Hof Method have been modulated to a scientifically reproducible mindset & physical training program for add-on therapy of axSpA. Specifically, it has been adjusted for potential functional limitations of axSpA.

Primary Objective: To investigate whether the add-on mindset & physical therapy program can safely be applied in patients with active axSpA using clinical safety parameters.

Secondary Objective: To assess whether the add-on mindset & physical therapy program can modulate objective signs of inflammation in patients with active axSpA using serum biomarkers (e.g. CRP).

Exploratory objective: To assess whether the add-on mindset & physical therapy program has an influence on the Ankylosing Spondylitis Disease Activity Score, quality of life, and depressive symptoms (HADS), and to explore the predictive role of generalized and specific outcome expectancies in patients with active axSpA

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of axSpA as assessed by the treating rheumatologist fulfilling the ASAS classification for axial SpA [Rudwaleit 2009]
* Between 18 and 45 years of age at screening
* Active disease as defined by an Ankylosing Spondylitis Disease Activity Score (ASDAS) of >2.1 and a CRP value of ≥5 at the screening visit.
* Ability and willingness to participate to the study and give written informed consent.

Exclusion Criteria:

* Patients who cannot give written consent or, in the opinion of the investigator, cannot comply to the requirements of the study protocol. Significant comorbidity, including a cardiac, renal, hepatic, neurological, metabolic or any other severe disease, which in the opinion of the investigator may interfere with the study or lead to deleterious effects for the patient.
* Recent history of (or persistent) infection requiring hospitalization or antibiotic treatment within 4 weeks of baseline.
* If female, patient should not be pregnant. A urine pregnancy-test will be performed at screening and has to be negative.
* Initiation of treatment with corticosteroids or DMARDs (synthetic and biologic) within 8 weeks before screening.
* Initiation of treatment with NSAID within 2 weeks before screening.
* Variation of the treatment doses within 6 weeks of screening.
* Intra-articular injection with corticosteroids within 4 weeks prior to screening.
* Daily doses of systemic corticosteroids exceeding the equivalent of 10 mg prednisolone per day.
* Use of other drugs and treatments that may affect the evaluation of systemic inflammation as judged by the investigator.
* Cardiovascular risk factors such as a personal history of cardiovascular disease, familial history of major adverse cardiovascular events (MACE) at age younger than 45 yrs, hypercholesterolemia and stroke.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-04-21 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 60 days
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment
Change in CRP value | 60 days

SECONDARY OUTCOMES:
Change in circulating cytokines | 30, 60, 180 days
Change in other serum inflammation biomarkers (ESR, calprotectin) | 30, 60, 180 days

OTHER OUTCOMES:
Change in disease activity as measured by the Ankylosing Spondylitis Disease Activity Score (ASDAS) | 30, 60, 180 days
Change in quality of life as measured by the SF-36 | 30, 60, 180 days
Change in quality of life as measured by the EQ-5D | 30, 60, 180 days
Change in depressive symptoms as measured by the Hospital Anxiety Depression Score (HADS). | 30, 60, 180 days
Generalized expectations as measured by the Eysenck Personality Questionnaire - Neuroticism scale (EPQ-N) | Baseline
Generalized expectations as measured by the Eysenck Personality Questionnaire - Life Orientation Test-Revised (LOT-R). | Baseline
Specific expectations regarding the effects of the training, measured by VAS scales that are framed to the specific intervention. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Baeten, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (2):
- Netherlands (2):
  - Academic Medical Center, Amsterdam
  - Ziekenhuis Bernhoven, Uden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kox M, Stoffels M, Smeekens SP, van Alfen N, Gomes M, Eijsvogels TM, Hopman MT, van der Hoeven JG, Netea MG, Pickkers P. The influence of concentration/meditation on autonomic nervous system activity and the innate immune response: a case study. Psychosom Med. 2012 Jun;74(5):489-94. doi: 10.1097/PSY.0b013e3182583c6d. PMID 22685240
- [Result] Kox M, van Eijk LT, Zwaag J, van den Wildenberg J, Sweep FC, van der Hoeven JG, Pickkers P. Voluntary activation of the sympathetic nervous system and attenuation of the innate immune response in humans. Proc Natl Acad Sci U S A. 2014 May 20;111(20):7379-84. doi: 10.1073/pnas.1322174111. Epub 2014 May 5. PMID 24799686
- [Derived] Buijze GA, De Jong HMY, Kox M, van de Sande MG, Van Schaardenburg D, Van Vugt RM, Popa CD, Pickkers P, Baeten DLP. An add-on training program involving breathing exercises, cold exposure, and meditation attenuates inflammation and disease activity in axial spondyloarthritis - A proof of concept trial. PLoS One. 2019 Dec 2;14(12):e0225749. doi: 10.1371/journal.pone.0225749. eCollection 2019. PMID 31790484